CLINICAL TRIAL: NCT03045614
Title: Prevalence and Predictors of Kidney Disease, and Long-Term Renal Outcome in Pulmonary Hypertension
Brief Title: Kidney Disease and Pulmonary Hypertension
Status: Completed | Type: Observational
Sponsor: University of Giessen (Other)
Responsible Party: Principal Investigator, Faeq Husain, Senior Physician Nephrology, University of Giessen
Other Study IDs: AZ 238/16
Record Dates: First submitted 2017-02-04; First posted 2017-02-07 (Estimated); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Collection of only residual material (blood, urine) for Deutsche Zentrum für Lungenforschung Biobank.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Evaluation of the prevalence of kidney disease, hemodynamic predictors and long-term renal outcome in patients with invasively diagnosed pulmonary hypertension.

DETAILED DESCRIPTION:
This study aims to determine the prevalence of kidney disease, hemodynamic predictors and long-term renal outcome of in-hospital patients with invasively diagnosed pulmonary hypertension at the Department of Pulmonology, University Hospital Giessen and Marburg, Giessen, Germany between 1999 and 2016.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years
* subjects with invasively diagnosed pulmonary hypertension at rest and available renal function and spot urine data at day of right heart catheterization between March 1999 and December 2016 at the Department of Pulmonology, University Hospital Giessen and Marburg, Giessen, Germany

Exclusion Criteria:

* subjects with estimated GFR <15ml/min/1.73m2 or prior dialysis
* pre-existing acute kidney injury
* non-end stage renal disease with extracorporeal or peritoneal ultrafiltration due to diuretic-resistant fluid overload
* primary kidney disease requiring active immunosuppression
* autosomal dominant polycystic kidney disease
* if subjects are pregnant
* if subjects are recipients of solid-organ transplants
* subjects with pulmonary hypertension with unclear/multifactorial mechanisms (WHO group 5 pulmonary hypertension)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with invasively diagnosed pulmonary hypertension between March 1999 and December 2016 at reference center for pulmonary hypertension, University Hospital Giessen, Germany.
Sampling Method: Non-Probability Sample
Enrollment: 824 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-08-27 (Actual); Study Completion 2018-08-28 (Actual)

PRIMARY OUTCOMES:
Changes in estimated glomerular filtration rate (GFR) in each class of pulmonary hypertension during follow-up period | 3 years follow-up
  Estimated GFR (Chronic Kidney Disease Epidemiology Collaboration) will be used over follow-up period to determine changes in renal function
Impact of renal function on deterioration of pulmonary hypertension during follow-up period | 3 years follow-up
  Changes in estimated GFR (Chronic Kidney Disease Epidemiology Collaboration) over follow-up period will be correlated with clinical worsening of pulmonary hypertension (as determined by echocardiography, 6-minute-walk, New York Heart Association classification, b-type natriuretic peptide)

SECONDARY OUTCOMES:
Impact of pulmonary hypertension-related morbidity on renal function decline | 3 years follow-up
  Severity of pulmonary hypertension (progress pulmonary hypertension, unscheduled hospitalization due to worsening of pulmonary hypertension, mortality) will be correlated with changes in renal function (as determined by estimated GFR [Chronic Kidney Disease Epidemiology Collaboration])
Prevalence of proteinuria in pulmonary hypertension | At baseline
  24 hours urine collection at baseline will be assessed to predict progress of pulmonary hypertension
Impact of pulmonary hypertension-specific therapy on renal function decline | 3 years follow-up
  Estimated GFR (Chronic Kidney Disease Epidemiology Collaboration) over follow-up period will be assessed to show association of pulmonary hypertension-specific therapy on renal function

CONTACTS AND LOCATIONS:
Overall Officials: Werner Seeger, MD, Study Director — University Clinic Giessen and Marburg, Campus Giessen
Locations (1):
- University Clinic Giessen and Marburg - Campus Giessen, Giessen, Hesse, Germany

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study are available from the corresponding author upon reasonable request.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Unlimited
Access Criteria: The data that support the findings of this study are available from the corresponding author upon reasonable request.

REFERENCES:
- [Result] Navaneethan SD, Wehbe E, Heresi GA, Gaur V, Minai OA, Arrigain S, Nally JV Jr, Schold JD, Rahman M, Dweik RA. Presence and outcomes of kidney disease in patients with pulmonary hypertension. Clin J Am Soc Nephrol. 2014 May;9(5):855-63. doi: 10.2215/CJN.10191013. Epub 2014 Feb 27. PMID 24578332
- [Result] Husain-Syed F, Slutsky AS, Ronco C. Lung-Kidney Cross-Talk in the Critically Ill Patient. Am J Respir Crit Care Med. 2016 Aug 15;194(4):402-14. doi: 10.1164/rccm.201602-0420CP. PMID 27337068